CLINICAL TRIAL: NCT00969852
Title: [11C] Sertraline PET Imaging Study That Investigates Pharmacokinetics and Pharmacodynamics of Sertraline After Low Dose Administration
Brief Title: Pharmacokinetics and Pharmacodynamics of Sertraline After Low Dose Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health, Welfare and Family Affairs (Unknown); Korea National Enterprise for Clinical Trials (Other)
Responsible Party: Kyung-Sang Yu/Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUCPT09_Sertraline
Record Dates: First submitted 2009-08-29; First posted 2009-09-01 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: Sertraline; PET; Serotonin receptor occupancy; PK-PD Model
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sertraline (Experimental): Single Arm
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Multiple doses of 5, 25, and 50 mg Sertraline for 6 days each period.
  Other Names: Zoloft(Pfizer)

SUMMARY:
This study aimed to explore the pharmacokinetics and pharmacodynamics of low dose sertraline with [11C] sertraline positron emission tomography (PET) study.

DETAILED DESCRIPTION:
Open, one arm, single sequence, 3-period, dose escalating study for healthy volunteers are investigated. Ten subjects may be enrolled.

Subjects receive baseline [11C] sertraline PET.

Period 1 Subjects receive 5 mg of sertraline every day. After 6 day of medication, pharmacokinetic and PET studies are performed.

Period 2 Subjects receive 25 mg of sertraline every day. After 6 day of medication, pharmacokinetic and PET studies are performed.

Period 3 Subjects receive 50 mg of sertraline every day. After 6 day of medication, pharmacokinetic and PET studies are performed.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 50 years of age, inclusive (age based on the date to give the informed consent)
* Weight: Over 55 kg, within ±20% of ideal body weight
* Subject who are reliable and willing to make themselves available during the study period, are willing to follow the study protocol, and give their written informed consent voluntarily

Exclusion Criteria:

* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease
* History of a significant surgical resection of gastrointestinal tract except appendectomy
* Abnormal clinical laboratory findings, especially for AST or ALT > 1.25 fold of upper normal limit
* Subject who has phobia for PET scan
* History or evidence of drug abuse
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any OTC medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (If used medication is considered acceptable by investigator, patients can be included)
* Participation in clinical trials of any drug within 2 months prior to the participation of the study
* Donation of whole blood within 2 months or a unit of blood within 1 month prior to the start of study
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Serotonin receptor occupancy | Day -1, Day 7, Day 14, Day 21

SECONDARY OUTCOMES:
Plasma concentration of sertraline | Day 4, 5, 6, 7, 11, 12, 13, 14, 18, 19, 20, 21

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin KH, Kim KP, Lim KS, Kim JW, Lee YS, Yang BY, Lee JS, Jung JM, Yoon SH, Jang IJ, Yu KS. A positron emission tomography microdosing study with sertraline in healthy volunteers. Int J Clin Pharmacol Ther. 2012 Mar;50(3):224-32. doi: 10.5414/cp201644. PMID 22373835